CLINICAL TRIAL: NCT00312793
Title: Phase 2 Study to Evaluate the Efficacy and Safety of Electronic Stimulation of the Quadriceps Muscle in the Thigh by the MyoSpare Device, in Patients Who Underwent Reconstruction of the Anterior Cruciate Ligament (ACL)
Brief Title: The Efficacy and Safety of Electronic Stimulation in Patients Who Underwent Reconstruction of the Anterior Cruciate Ligament
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: the study stopped becaust the sponsor did not wish to proceede with the study
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST02-HMO-CTIL
Record Dates: First submitted 2006-04-10; First posted 2006-04-11 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Knee Injuries
Keywords: Anterior Cruciate Ligament reconstruction surgery
MeSH Terms: conditions — Knee Injuries

INTERVENTIONS:
Device: stimulation of the quadriceps muscle with Myospare

SUMMARY:
This study is designed to evaluate the efficacy and safety of Myospare, a non-invasive device, which is connected to the body via electrodes placed in the injured leg. The electrodes which are placed in the middle or upper thigh will stimulate the quadriceps muscle.

Myospare will be installed 1 day after the anterior cruciate ligament (ACL) reconstruction surgery and will be removed after 6 weeks of treatment. The patients will be assigned to two groups:

1. Physiotherapy plus Myospare
2. Only physiotherapy

The hypothesis of the study is that electrical stimulation combined with voluntary exercise is more effective than voluntary exercise alone.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18-40 years old.
2. Subjects who are planning to undergo ACL surgery.
3. The surgery is performed within 3 weeks - 5 years since the injury.
4. Ability to follow instructions during the study period.
5. Signed Informed Consent.

Exclusion Criteria:

1. Bi-lateral surgery of the knee
2. Recurrent ACL surgery (patients who already underwent ACL surgery)
3. Complex injuries (a combination of posterior and anterior cruciate and lateral ligament injury)
4. Patients who underwent or are planned to undergo cartilage implantation.
5. Patients who underwent or are planned to undergo meniscus stitching.
6. Additional fracture/s in the lower limbs as a result of the same injury.
7. Signs of infection in the surgical wounds while installing the Myospare device.
8. Known skin hypersensitivity.
9. Known heart disease
10. Patients with a cardiac pacemaker.
11. History of peripheral blood vessel disease
12. Administration of drugs which might disrupt bone metabolism:

    * Total accumulating dosage of 150 gr' prednisone or any other glucocorticoid for seven days or more, within 6 months prior to the trial.
    * Calcitonin for 7 days or more, within 6 months prior to the trial.
    * Bisphosphonates for 30 days or more within 12 months prior to the study.
    * Fluoride for bone strengthening for 30 days or more within 12 months prior to the study.
    * Vitamin D or vitamin D metabolite for bone strengthening for 30 days or more within 12 months prior to the study.
    * Current treatment with chemotherapeutic drugs.
13. Past or current malignant disease within 10 years of study entry.
14. Participating in another clinical study during the past four weeks.
15. Patients who are planned to undergo femoral nerve block.
16. Patients claiming social security/work accident benefits.
17. Professional athletes whose livelihood depends on sports.
18. Pregnant and or lactating women.
19. Additional symptoms, which in the doctor's opinion would prevent inclusion of the patient in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)

PRIMARY OUTCOMES:
the outcome measure is muscle weakness and atrophy (after six weeks) measured by isometric device

SECONDARY OUTCOMES:
range of movement measured by protractor
swelling measure by physical examination
stability of the knee measure by KT1000
knee history measure by IKDC2000
functional preservation measure by single hop tests and triple hop tests

CONTACTS AND LOCATIONS:
Overall Officials: Meir Libergall, Prof., Principal Investigator — Hadassah Medical Organization; Joseph Lowe, Dr., Study Director — Hadassah Medical Organization; Adi Fridman, Dr., Study Chair — Hadassah Medical Organization; Naama Constantini, Dr., Study Chair — Hadassah Medical Organization; Gabi Agar, Dr., Study Director — Asaf Ha'rofe Medical Organization; Yiftah Bar, Dr., Study Chair — Asaf Ha'rofe Medical Organization; Gideon Man, Dr., Study Director — Meir Medical Organization; Yiftah Hetzroni, Dr., Study Chair — Meir Medical Organization
Locations (3):
- Israel (3):
  - Asaf Ha'rofe Orthopedic Department, Beer Yaacov
  - Hadassah Orthopedic Department, Jerusalem
  - Meir Orthopedic Department, Kfar Saba